CLINICAL TRIAL: NCT02679365
Title: Double Lock Versus Continuous Non-locking Technique for Closure of Rectus Sheath in Cesarean Sections on Post-operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, dr mohammed elsafty, Associate Professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2476ASU
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- group a (Experimental): This arm will have lower segment cesarean section done with double locking technique for closure of Rectus Sheath.
  Interventions: Procedure: lower segment cesarean section and double lock closure of rectus sheath
- group b (Active Comparator): This arm will have lower segment cesarean section done with continuous non-locking technique for closure of rectus sheath.
  Interventions: Procedure: lower segment cesarean section and continuous non-locking closure of rectus sheath

INTERVENTIONS:
Procedure: lower segment cesarean section and double lock closure of rectus sheath
  Arms: group a
Procedure: lower segment cesarean section and continuous non-locking closure of rectus sheath
  Arms: group b

SUMMARY:
In this trial we compare the effect of 2 closure techniques of the rectus sheath during cesarean sections on postoperative pain. One closure technique is double lock technique and the other is the conventional continuous non-locking technique.

ELIGIBILITY:
Inclusion Criteria:

* first cesarean section

Exclusion Criteria:

* urgent cesarean section
* previous abdominal surgery
* previous cesarean section
* obstetric and medical complications

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
postoperative pain evaluated by VAS | first week postoperative

SECONDARY OUTCOMES:
operative time | intraoperative